CLINICAL TRIAL: NCT07060872
Title: A Randomized Controlled Interventional Study on the Effects of Spirulina Supplementation on Anxiety in Children With Non-Idiopathic Autism
Brief Title: the Effect of Formulation on Anxiety in Autist Childre A Randomized Controlled Trial Assesses Spirulina Syrup Plus Risperidone in Children With Non-idiopathic Autism. Anxiety is Measured Using the SCAS (Parent Version) Via Daily Online Surveys for One Week and Throughout a 3-month Follow-up Period.
Acronym: Autism Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Sadoughi University of Medical Sciences and Health Services (Other)
Responsible Party: Principal Investigator, Sanaz Alamdar, Graduate Student, Shahid Sadoughi University of Medical Sciences and Health Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.SSU.REC
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Age 3 to 7 Years; Mild Autism Spectrum; no Other Illness or Disorder
Keywords: Autism; Anxiety; Spirulina; Pharmaceutical supplement
MeSH Terms: conditions — Autistic Disorder; Anxiety Disorders | interventions — Risperidone

STUDY DESIGN:
Intervention Model Description: A group of 41 people took the formulation and a group of 41 people took a placebo
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spirulina Syrup (Experimental): * Spirulina Syrup
  * Risperidone
  Interventions: Dietary Supplement: Spirulina Syrup; Drug: Risperidone
- Placebo Syrup (Placebo Comparator): * Placebo Syrup
  * Risperidone
  Interventions: Dietary Supplement: Placebo Syrup; Drug: Risperidone

INTERVENTIONS:
Dietary Supplement: Spirulina Syrup — A natural dietary supplement derived from Spirulina algae, administered orally as a syrup formulation. Used as an adjunct therapy to assess its potential effect on reducing anxiety symptoms in children with non-idiopathic autism. Dosage and duration are standardized according to study protocol.
  Arms: Spirulina Syrup
Dietary Supplement: Placebo Syrup — Placebo Syrup
  Arms: Placebo Syrup
Drug: Risperidone — Risperidone

SUMMARY:
The aim of this study is to evaluate the effect of a Spirulina syrup formulation on reducing anxiety in children with non-idiopathic autism. Participants are referred to a private clinic and assessed by a pediatric neurology subspecialist to confirm the diagnosis. Informed consent is obtained from the parents. Patients are randomly assigned to two groups. The intervention group receives standard treatment (Risperidone tablets) plus Spirulina syrup, while the control group receives Risperidone plus a placebo. Anxiety is measured using the parent version of the Spence Children's Anxiety Scale (SCAS), which includes 38 items rated on a 4-point Likert scale. The questionnaire is administered online via the Porsline platform, and links are sent nightly via social media starting before treatment and continuing daily for one week after treatment initiation, then regularly over a 3-month follow-up period. Data will be analyzed using SPSS version 16. The SCAS consists of six subscales: separation anxiety, social anxiety, phobia, generalized anxiety, panic, and obsessive-compulsive symptoms.

DETAILED DESCRIPTION:
Detailed Description

Autism Spectrum Disorder (ASD) is a neurodevelopmental condition characterized by persistent challenges in social interaction, communication, and restricted, repetitive patterns of behavior, interests, or activities. According to the latest data from the U.S. Centers for Disease Control and Prevention (CDC), approximately 1 in 54 children aged 8 years is diagnosed with ASD. The exact etiology of ASD remains unclear, but both genetic and environmental risk factors-including advanced parental age, prenatal infections, and complications during pregnancy-have been implicated.

ASD presents with a heterogeneous range of symptoms and severity. Some children may demonstrate intellectual disability, language delays, sensory sensitivities, stereotyped behaviors, and resistance to change. Others may show above-average intelligence, articulate speech, and creative talents. In addition to core symptoms, individuals with ASD often suffer from comorbidities such as anxiety, depression, gastrointestinal disturbances, and sleep problems. These comorbid conditions can significantly impair quality of life and increase the burden on families, necessitating a multidisciplinary treatment approach.

While no definitive cure for ASD currently exists, evidence-based interventions such as behavioral therapies, educational programs, and pharmacological treatments aim to manage core symptoms and associated conditions. Common pharmacologic interventions include antipsychotic medications such as risperidone to manage irritability and aggression. However, these medications often come with undesirable side effects. Consequently, there is a growing interest in complementary and alternative medicine (CAM) to support children with ASD.

Recent studies suggest that 50-95% of families with ASD-affected children explore CAM therapies, including herbal medicine, dietary supplements, and special diets. Despite limited empirical evidence, several traditional remedies have shown promise in mitigating symptoms or improving physiological functions in ASD.

In this clinical trial, we evaluate the potential anxiolytic effects of Spirulina syrup and Lemon Verbena (Lippia citriodora) syrup in children with non-idiopathic ASD. Participants are recruited from a private pediatric neurology clinic. All children are diagnosed by a pediatric neurology subspecialist, and parental informed consent is obtained before inclusion. Participants are randomized into two groups. The intervention group receives Spirulina syrup in addition to standard treatment with risperidone tablets, while the control group receives a placebo syrup with standard risperidone therapy.

Anxiety levels are measured using the Spence Children's Anxiety Scale - Parent Version (SCAS-P), which includes 38 items rated on a 4-point Likert scale (0 = never, 3 = always). This scale evaluates six subdomains: separation anxiety, social phobia, specific phobia, generalized anxiety, panic/agoraphobia, and obsessive-compulsive symptoms. The SCAS questionnaire is administered daily via the Porsline online platform. A secure link is shared with parents through social media from the week prior to intervention and continues nightly for one week after initiation. Responses are collected regularly throughout the 3-month follow-up period. Data will be analyzed using SPSS version 16.

Moreover, to evaluate the potential effectiveness of Spirulina syrup and lemon verbena (Lippia citriodora) extract in improving symptoms of Autism Spectrum Disorder (ASD), particularly in reducing anxiety symptoms, a randomized, placebo-controlled clinical trial was designed. The intervention is administered in combination with standard pharmacological therapy (Risperidone tablets) in a population of pediatric patients diagnosed with non-idiopathic autism.

This clinical study enrolls participants from a private clinic where children referred for ASD concerns are assessed by a pediatric neurology subspecialist. Inclusion criteria include children formally diagnosed with non-idiopathic ASD. After obtaining informed consent from parents, the children are randomly assigned to two groups: an intervention group receiving standard care with Risperidone and Spirulina syrup, and a control group receiving standard care with a placebo syrup.

The main outcome measure in this study is the level of anxiety, assessed using the Spence Children's Anxiety Scale (SCAS) - Parent Version. This scale consists of 38 items distributed across six subscales: separation anxiety, social anxiety, obsessive-compulsive symptoms, panic/agoraphobia, generalized anxiety, and fears of physical injury. Parents complete the SCAS via an online platform (Porsline) daily starting one week before treatment and continuing for three months following treatment initiation.

The anticipated therapeutic benefits of Spirulina and lemon verbena stem from their biochemical properties. Spirulina, a blue-green algae (Arthrospira maxima), is rich in protein, vitamins, antioxidants, and anti-inflammatory compounds. It may enhance immune function, reduce systemic inflammation, and improve oxidative stress, all of which are potentially implicated in the pathophysiology of ASD. Additionally, Spirulina has been studied for its anxiolytic effects and its potential to support cognitive performance.

Lemon verbena, a medicinal plant known for its calming effects, is traditionally used for its anxiolytic, anti-inflammatory, and digestive benefits. Bioactive compounds found in lemon verbena, such as flavonoids and phenolic acids, have demonstrated significant antioxidant and anti-inflammatory activity in prior in vitro and in vivo studies. These properties may offer additional support in addressing anxiety and gastrointestinal issues frequently seen in children with ASD.

Safety assessments include monitoring adverse events and routine clinical evaluations. Data analysis is performed using SPSS version 16. Descriptive statistics, repeated-measures ANOVA, and post-hoc tests will assess within- and between-group changes over time. The primary hypothesis is that children in the intervention group will show statistically significant reductions in anxiety symptoms compared to the control group.

This study contributes to the growing body of research into complementary and alternative medicine (CAM) approaches for ASD management. While no definitive cure for ASD currently exists, integrating safe and potentially effective natural compounds like Spirulina and lemon verbena into treatment protocols may offer additional benefits for improving the quality of life of children with ASD and their families.

Further research is warranted to validate the efficacy, safety, and mechanisms of action of these natural supplements. Should the outcomes of this clinical trial prove promising, they may lay the foundation for larger, multicenter trials and pave the way for evidence-based integration of traditional medicine with conventional ASD care practices.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with non-idiopathic autism, confirmed by a pediatric neurology subspecialist

  * Age range: [3 to 7 years]
  * Parental informed consent obtained
  * Ability to complete online anxiety questionnaires with parental assistance

Exclusion Criteria:

* • Presence of other major neurological or psychiatric disorders

  * Known allergy or intolerance to Spirulina or Risperidone
  * Participation in other clinical trials within the past 3 months
  * Severe medical conditions that contraindicate the use of study medications

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety symptoms based on the Spence Children's Anxiety Scale (Parent Version) total score | From baseline to 3 months after treatment initiation
  Anxiety symptoms will be assessed using the Spence Children's Anxiety Scale (SCAS) - Parent Version, a 38-item validated tool. Total score changes will be used to evaluate treatment efficacy.

SECONDARY OUTCOMES:
Change in subscale scores of SCAS (e.g., separation anxiety, social anxiety, generalized anxiety, etc.) | From baseline to 3 months after treatment initiation
  SCAS subscale scores will be analyzed to determine which domains of anxiety are most affected by Spirulina supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanaz Alamdar, Yazd, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://revmov.miencocienanco.1oero.cou.co/ordc/e/view/coc